CLINICAL TRIAL: NCT00318110
Title: Multicenter Phase II Study of Non-Myeloablative Allogeneic Stem Cell Transplantation Using Matched Unrelated Donor for Metastatic Renal Cell Carcinoma
Brief Title: Matched Unrelated Donor Transplant for Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to meet subject enrollment goal.
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T00008; NCT00429130 (obsolete NCT alias)
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic; Renal; Cell; Carcinoma; Unrelated; Donor; Transplant; stage IV; clear cell
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MUD treatment (Experimental): NST using MUD for metastatic renal cell carcinoma
  Interventions: Procedure: NST using MUD for metastatic renal cell carcinoma

INTERVENTIONS:
Procedure: NST using MUD for metastatic renal cell carcinoma — Preparative regimen:
  Fludarabine 25 mg/m2 IV once a day x 5 days (-6,-5,-4,-3,-2) Melphalan 70 mg/m2 IV once a day x 2 days (-3,-2) Donor Stem Cell Infusion: Stem cells will be infused on day 0 GVHD prophylaxis: Tacrolimus and methotrexate 5 mg/m2 IV day 1, 3, 6 and 11

SUMMARY:
The purpose of this study is to find out what effects (good and bad) a stem cell transplant from an unrelated donor will have for patients with kidney cancer that has spread to other parts of the body (metastasized).

DETAILED DESCRIPTION:
Standard treatment for kidney cancer that has spread to other parts of the body may include immunotherapy (a therapy that uses the body's natural immune system to fight cancer) and cytokines (proteins found in the body). If these treatments are not successful at controlling the cancer then chemotherapy or thalidomide are used. Chemotherapy and thalidomide will not cure kidney cancer but they may control the disease in some patients.

In some patients, transplants are now proposed for study. Stem cells (from bone marrow or the bloodstream) are normally used to treat cancers of the blood, not kidney cancer. Since researchers are still learning about using stem cell transplants for kidney cancer, the study is considered a research study. Patients participating in this study will receive smaller doses of chemotherapy drugs to prepare them for the transplant than patients who have a standard transplant. This type of transplant is called a "reduced intensity" transplant. A reduced intensity transplant uses the cell-killing activity of the transplanted donor stem cells to attack the recipient's cancer cells. This is called graft-versus-tumor-effect (GVT). Previous studies have shown that GVT may be greater if the donor is not related to the recipient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic (stage IV) renal cell carcinoma (RCC) predominately clear cell type
* Prior nephrectomy
* Available HLA-matched (8/8, 7/8) unrelated donor
* At least one prior immunotherapy; or immunotherapy + chemotherapy; or targeted therapy, for metastatic RCC.
* Adequate organ function

Exclusion Criteria:

* Prior allogeneic stem cell transplantation
* RCC with histology other than clear cell type
* History or presence of brain metastasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Determine the best rate of tumor response of complete response (CR) + complete unconfirmed response (CRU) + partial response (PR) within 6 months after matched unrelated donor (MUD) nonmyeloablative stem cell transplantation (NST) | 6 months

SECONDARY OUTCOMES:
Overall survival after MUD NST | Two years
Rate of complete donor myeloid and lymphoid chimerism after MUD NST | One year
Incidence and severity of acute and chronic graft-versus-host disease (GvHD) after MUD NST | Two years
Incidence of treatment-related mortality (TRM) | 100 Days
Assess cytotoxic T-lymphocyte reactivity | One year
Assess antibody activity against potential tumor antigenic peptides in graft-versus-renal cell carcinoma (RCC) effect | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, M.D., Ph.D., Study Chair — MDACC
Locations (5):
- United States (5):
  - University of California - Los Angeles, Los Angeles, California
  - Shands - University of Florida, Gainesville, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Only 2 subjects enrolled prior to study closure due to slow accrual.

REFERENCES:
- See also: Click for more information about the Center for International Blood and Marrow Transplant Research — http://www.CIBMTR.org